CLINICAL TRIAL: NCT01567163
Title: A Study to Evaluate the Potential of Concomitant Ramucirumab to Affect the Pharmacokinetics of Docetaxel in Patients With Advanced Malignant Solid Tumors
Brief Title: A Study of Ramucirumab and Docetaxel in Participants With Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14434; CP12-0713 (Other: ImClone Systems); I4T-IE-JVCC (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-03-28; First posted 2012-03-30 (Estimated); Results first posted 2014-06-18 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Malignant Solid Tumor
Keywords: Advanced Malignant Solid Tumors
MeSH Terms: interventions — Ramucirumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ramucirumab (IMC-1121B) and docetaxel (Experimental): Cycle 1: docetaxel administered on Day 1 of 3-week cycle
  Cycle 2: ramucirumab and docetaxel administered on Day 1 of 3-week cycle
  Cycle 3 and beyond: ramucirumab and docetaxel administered on Day 1 of each 3-week cycle
  Extension Phase: ramucirumab and docetaxel administered on Day 1 of each 3-week cycle
  Interventions: Biological: Ramucirumab; Drug: Docetaxel

INTERVENTIONS:
Biological: Ramucirumab — ramucirumab 10 milligrams/kilogram (mg/kg) intravenous infusion, administered on Day 1 of 3-week cycle
  Other Names: IMC-1121B; LY3009806
Drug: Docetaxel — docetaxel 75 milligrams/square meter (mg/m^2) intravenous infusion administered on Day 1 of each 3-week cycle

SUMMARY:
The purpose of this study is to assess the effect of concomitant ramucirumab on the pharmacokinetics of docetaxel in participants with advanced malignant solid tumors.

Participants who do not complete both Cycle 1, Day 1, and Cycle 2, Day 1 according to schedule will be replaced for the purpose of analysis; these participants may continue to receive study therapy. No dose reductions, delayed or missed doses are allowed during Cycles 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

* Participant has histologic or cytologic documentation of a malignant solid tumor
* Participant has an advanced solid tumor that is resistant to standard therapy or for which no standard therapy is available
* Participant has had 0-1 prior taxane-containing treatment regimens (including taxane monotherapy), which must have been completed at least 6 months before the first dose of study medication. Prior bevacizumab is allowed.
* Participant has resolution to Grade ≤ 1 (except where otherwise stated in this eligibility criteria) by the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 4.0 (NCI-CTCAE v 4.0) of all clinically significant toxic effects of prior chemotherapy, surgery, radiotherapy, or hormonal therapy
* Participant has an Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0-2
* Participant has adequate hematologic function (absolute neutrophil count [ANC] ≥ 1500 cells/liter (cells/L), hemoglobin ≥ 10 grams/deciliter (g/dL), and platelet count ≥ 100,000 cells/microliter (cells/mcL)]. Blood transfusion is allowed but must be completed 48 hours before study drug administration.
* Participant has adequate hepatic function (bilirubin ≤ 1.5 times the upper limit of normal [x ULN], aspartate transaminase [AST] and alanine transaminase [ALT] ≤ 1.5 x ULN)
* Participant has serum creatinine ≤ 1.5 x ULN. If serum creatinine > 1.5 x ULN, the calculated creatinine clearance [CrCl] should be ≥ 40 milliliters/minute (mL/min)
* Participant's urinary protein is <2+ on dipstick or routine urinalysis (UA) at study entry
* Participant must have adequate coagulation function as defined by an international normalized ratio (INR) of ≤ 1.5 and a partial thromboplastin time (PTT) or an activated PTT (aPTT) ≤ 1.5 x ULN
* Women with childbearing potential must have a negative serum or urine pregnancy test. Eligible participants of reproductive potential (both sexes) agree to use adequate method of contraception during the study period and for 12 weeks after the last dose of study medication.

Exclusion Criteria:

* Has a known allergy or hypersensitivity to any of the treatment components
* Are currently enrolled in, or discontinued within the last 14 days from, a clinical trial involving an investigational product or non-approved use of a drug or device, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Has received a therapeutic monoclonal antibody within 42 days prior to first dose of study medication
* Has received radiotherapy within 14 days prior to first dose of study medication
* Has received cytotoxic chemotherapy within 21 days prior to first dose of study medication
* Is receiving concurrent treatment with another anticancer therapy, including chemotherapy, immunotherapy, hormonal therapy (except for androgen deprivation therapy for prostate cancer), radiation therapy, chemoembolization, targeted or other investigational anticancer therapy
* Is receiving chronic therapy with nonsteroidal anti-inflammatory agents or other antiplatelet agents. (Aspirin use at doses up to 325 milligrams/day (mg/day) and analgesic agents with no or low bleeding risk are permitted.)
* Has a history of uncontrolled hereditary or acquired bleeding or thromboembolic disorders
* Has experienced any arterial thromboembolic event, including myocardial infarction (MI), unstable angina, stroke or transient ischemic attack (TIA), within 6 months prior to first dose of study medication
* Has a history of deep vein thrombosis, pulmonary embolism, or any other significant thromboembolism during the 3 months prior to first dose of study medication
* Has experienced a Grade 3 or 4 hemorrhagic event within 3 months prior to first dose of study medication
* Has experienced peripheral neuropathy ≥ Grade 2 at any time prior to study entry
* Has a bowel obstruction, history or presence of inflammatory enteropathy or extensive intestinal resection, Crohn's disease, ulcerative colitis, or chronic diarrhea
* History of gastrointestinal perforation and/or fistulae within 6 months prior to randomization
* Has an ongoing or active infection requiring treatment with intravenous antibiotics
* Has a serious or nonhealing wound, peptic ulcer, or bone fracture within 28 days prior to first dose of study medication
* Has uncontrolled hypertension despite standard medical management
* Has symptomatic congestive heart failure, symptomatic or poorly controlled cardiac arrhythmia, or any other serious, uncontrolled medical disorders, which in the opinion of the investigator would make the participant ineligible for participation in the study
* Has known brain or leptomeningeal metastases
* Has known positive status for human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome-related illness
* Has known active drug or alcohol abuse
* Has pulmonary lymphangitic involvement that results in pulmonary dysfunction requiring active treatment, including the use of oxygen
* Has had major surgery within 28 days prior to first dose of study medication or subcutaneous venous access device implantation within 7 days prior to first dose of study medication
* Has an elective or planned major surgery during the course of the trial
* If the primary cancer is non-small-cell lung cancer (NSCLC), there is radiographic evidence of intratumor cavitation, major blood vessel invasion or encasement by cancer, or proximity of cancer to major airways
* Has received prior ramucirumab (IMC-1121B) therapy
* Is receiving concomitant therapy with clinically relevant inhibitors or inducers of cytochrome P450 3A4 and 3A5 and/or isoenzymes
* Has cirrhosis at a level of Child-Pugh B (or worse), or cirrhosis and a history of hepatic encephalopathy, or ascites resulting from cirrhosis and requiring ongoing treatment with diuretics and/or paracentesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-07; Primary Completion 2012-12 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (6):
- United States (6):
  - ImClone Investigational Site, Ann Arbor, Michigan
  - ImClone Investigational Site, Detroit, Michigan
  - ImClone Investigational Site, New Brunswick, New Jersey
  - ImClone Investigational Site, Huntersville, North Carolina
  - ImClone Investigational Site, Cleveland, Ohio
  - ImClone Investigational Site, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Cycle 1: docetaxel 75-milligrams/square meter (mg/m^2) intravenous infusion administered on Day 1 of 3-week cycle
  Cycle 2: ramucirumab 10-milligrams/kilogram (mg/kg) intravenous infusion, followed by docetaxel 75-mg/m^2 intravenous infusion administered on Day 1 of 3-week cycle
  Cycle 3 and beyond: ramucirumab and docetaxel administered on Day 1 of each 3-week cycle
Period: Overall Study
Arm/Group | All Participants
Started | 22
Received at Least 1 Dose of Study Drug | 22
Drug-Drug Interaction Population | 18 (Completed Cycle 1, Day 1 and Cycle 2, Day 1 treatment with required assessments.)
Completed | 18
Not Completed | 4
Not completed — Progressive Disease | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of ramucirumab or docetaxel.
Arm/Group | All Participants
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 4
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Dose-Normalized Area Under the Concentration Versus Time Curve of Docetaxel From Time Zero to Infinity [AUC(0-∞)] Following a Single Dose in Cycle 1
Time Frame: Cycle 1: 0, 1, 1.5, 2, 3, 5, 7, 24, 48 and 72 hours post docetaxel infusion
Population: All participants who completed Cycle 1, Day 1 and Cycle 2, Day 1 treatment and had sufficient concentration data to calculate docetaxel AUC(0-∞) in Cycle 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour/milliliter/milligram
Groups:
- Docetaxel (Cycle 1): Cycle 1: docetaxel 75-milligrams/square meter (mg/m^2) intravenous infusion administered on Day 1 of 3-week cycle
Arm/Group | Docetaxel (Cycle 1)
Number analyzed (Participants) | 17
nanograms*hour/milliliter/milligram | 13.7 (40)

2. Primary Outcome: Pharmacokinetics: Dose-Normalized Area Under the Concentration Versus Time Curve of Docetaxel From Time Zero to Infinity [AUC(0-∞)] Following a Single Dose in Cycle 2
Time Frame: Cycle 2: 0, 1, 1.5, 2, 3, 5, 7, 24, 48 and 72 hours post docetaxel infusion
Population: All participants who completed Cycle 1, Day 1 and Cycle 2, Day 1 treatment and had sufficient concentration data to calculate docetaxel AUC(0-∞) in Cycle 2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour/milliliter/milligram
Groups:
- Docetaxel (Cycle 2): Cycle 2: ramucirumab 10-milligrams/kilogram (mg/kg) intravenous infusion and followed by docetaxel 75-milligrams/square meter (mg/m^2) intravenous infusion administered on Day 1 of 3-week cycle
Arm/Group | Docetaxel (Cycle 2)
Number analyzed (Participants) | 16
nanograms*hour/milliliter/milligram | 12.8 (30)
Statistical Analysis 1: Comparison: Docetaxel (Cycle 2); Test type: Superiority or Other; Mixed Models Analysis; Ratio geometric least squares (LS) means = 0.97, 90% CI 2-sided [0.84 to 1.10] — The ratio of geometric LS means was calculated using a mixed effect model adjusted for cycle, participant and random error. Ratio of geometric LS means is AUC(0-∞) of Cycle 2/Cycle 1

3. Primary Outcome: Pharmacokinetics: Dose-Normalized Maximum Observed Drug Concentration (Cmax) of Docetaxel in Cycle 1
Time Frame: Cycle 1: 0, 1, 1.5, 2, 3, 5, 7, 24, 48, and 72 hours post docetaxel infusion
Population: All participants who completed Cycle 1, Day 1 and Cycle 2, Day 1 treatment and had sufficient concentration data to calculate docetaxel Cmax in Cycle 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter/milligram
Arm/Group | Docetaxel (Cycle 1)
Number analyzed (Participants) | 17
nanograms/milliliter/milligram | 7.66 (76)

4. Primary Outcome: Pharmacokinetics: Dose-Normalized Maximum Observed Drug Concentration (Cmax) of Docetaxel in Cycle 2
Time Frame: Cycle 2: 0, 1, 1.5, 2, 3, 5, 7, 24, 48 and 72 hours post docetaxel infusion
Population: All participants who completed Cycle 1, Day 1 and Cycle 2, Day 1 treatment and had sufficient concentration data to calculate docetaxel Cmax in Cycle 2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter/milligram
Groups:
- Docetaxel (Cycle 2): Cycle 2: ramucirumab 10-milligrams/kilogram (mg/kg) intravenous infusion, followed by docetaxel 75-milligrams/square meter (mg/m^2) intravenous infusion administered on Day 1 of 3-week cycle
Arm/Group | Docetaxel (Cycle 2)
Number analyzed (Participants) | 17
nanograms/milliliter/milligram | 8.78 (37)
Statistical Analysis 1: Comparison: Docetaxel (Cycle 2); Test type: Superiority or Other; Mixed Models Analysis; Ratio of geometric least squares means = 1.14, 90% CI 2-sided [0.84 to 1.55] — The ratio of geometric least squares means was calculated using a mixed effect model adjusted for cycle, participant and random error. Ratio of Geo LS mean is Cmax of Cycle 2/Cycle 1

5. Secondary Outcome: Number of Participants With Treatment-Emergent Anti-Ramucirumab Antibodies
Description: Participants with treatment-emergent anti-ramucirumab antibodies were participants with a 4-fold increase (2 dilution increase) in immunogenicity titer over baseline titer, or participants who tested negative at baseline and positive post-baseline (at titer of ≥1:20).
Time Frame: Cycle 1, Day 1 through Cycle 2, Day 1 and 30 days after last dose of study drug
Population: All participants who completed Cycle 1, Day 1 and Cycle 2, Day 1 treatment who had immunogenicity samples collected at the specified time points.
Measure: Number; unit: participants
Arm/Group | All Participants
Number analyzed (Participants) | 17
participants
  Immunogenicity During Study (n=17) | 0
  Immunogenicity Post-Treatment (n=5) | 0

6. Secondary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve of Ramucirumab From Time Zero to Infinity [AUC(0-∞)] in the Presence of Docetaxel
Time Frame: Cycle 2: 1 hour prior to ramucirumab infusion, 0, 1, 2, 2.5, 3, 4, 6, 8, 25, 49, 73, 169, 265 and 337 hours post ramucirumab infusion
Population: All enrolled participants who received ramucirumab and had sufficient concentration data to calculate ramucirumab AUC(0-∞) in Cycle 2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*hour/milliliter (mcg*h/mL)
Groups:
- Ramucirumab: Cycle 2: ramucirumab 10-milligrams/kilogram (mg/kg) intravenous infusion, followed by docetaxel 75-milligrams/square meter (mg/m^2) intravenous infusion administered on Day 1 of 3-week cycle
Arm/Group | Ramucirumab
Number analyzed (Participants) | 11
micrograms*hour/milliliter (mcg*h/mL) | 42400 (32)

7. Secondary Outcome: Pharmacokinetics: Maximum Observed Drug Concentration (Cmax) of Ramucirumab in the Presence of Docetaxel
Time Frame: as for outcome 6
Population: All enrolled participants who received ramucirumab and had sufficient concentration data to calculate ramucirumab Cmax in Cycle 2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/milliliter (mcg/mL)
Groups:
- Ramucirumab: Cycle 2: ramucirumab 10-milligrams/kilogram (mg/kg) intravenous infusion and followed by docetaxel 75-milligrams/square meter (mg/m^2) intravenous infusion administered on Day 1 of 3-week cycle
Arm/Group | Ramucirumab
Number analyzed (Participants) | 18
micrograms/milliliter (mcg/mL) | 303.6 (28)

ADVERSE EVENTS:
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 11/22
Other Adverse Events (participants affected / at risk) | 20/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=22)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (2)
Clostridium difficile infection (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Wound infection (Infections and infestations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Nervous system disorder (Nervous system disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (4)
Embolism (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | All Participants (N=22)
Anaemia (Blood and lymphatic system disorders) | 6 (11)
Neutropenia (Blood and lymphatic system disorders) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 4 (8)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 12 (13)
Oral pain (Gastrointestinal disorders) | 3 (3)
Stomatitis (Gastrointestinal disorders) | 3 (5)
Vomiting (Gastrointestinal disorders) | 2 (2)
Asthenia (General disorders) | 2 (3)
Chest discomfort (General disorders) | 4 (4)
Chills (General disorders) | 2 (2)
Fatigue (General disorders) | 9 (15)
Oedema peripheral (General disorders) | 2 (4)
Pain (General disorders) | 2 (2)
Vulvovaginal mycotic infection (Infections and infestations) | 1/9 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 4 (7)
White blood cell count decreased (Investigations) | 9 (15)
Decreased appetite (Metabolism and nutrition disorders) | 5 (7)
Dehydration (Metabolism and nutrition disorders) | 2 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 6 (6)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (7)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 5 (7)
Headache (Nervous system disorders) | 4 (4)
Neuropathy peripheral (Nervous system disorders) | 3 (4)
Insomnia (Psychiatric disorders) | 2 (2)
Vaginal haemorrhage (Reproductive system and breast disorders) | 2/9 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (9)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5)
Nail discolouration (Skin and subcutaneous tissue disorders) | 2 (2)
Nail disorder (Skin and subcutaneous tissue disorders) | 2 (3)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 3 (4)
Hypertension (Vascular disorders) | 7 (8)
Hypotension (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed to delay independently publishing or disclosing data, findings or conclusions from the study except as part of a multi-center publication. Upon study publication or if the draft publication is not produced within approximately 6 months of the final report of the study results, investigators may independently publish, subject to confidential information review/redaction by sponsor. The sponsor may request publication delay up to 90 days to seek patent protection.